CLINICAL TRIAL: NCT02501447
Title: Feasibility of a Stress Reduction Intervention Study in Sickle Cell Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Miriam O. Ezenwa, Assistant Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Protocol # 2012-1084
Record Dates: First submitted 2015-07-13; First posted 2015-07-17 (Estimated); Last update posted 2015-07-17 (Estimated); Status verified 2015-07

CONDITIONS: Sickle Cell Disease; Stress
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Guided audio-visual relaxation group (Experimental): The guided relaxation (GR) intervention included a single 12-min GR video clip we administered to subjects at the baseline visit to determine the immediate effects of GR on stress and pain. The GR intervention also included six video clips, which ranged from 2 to 20 minutes in length to determine the short-term (2-week) effects of GR on stress and pain.
  Interventions: Behavioral: Guided audio-visual relaxation
- Attention Control group (No Intervention): For the attention control group, subjects engaged in a 12-min computer-based discussion about their sickle cell disease (SCD) experience. The audio-taped questions and onscreen directions were programmed for self-administration. Subjects' responses were captured via the microphone so that Data Collectors were not involved in this discussion process, and it was equivalent to the guided relation activity.

INTERVENTIONS:
Behavioral: Guided audio-visual relaxation
  Arms: Guided audio-visual relaxation group

SUMMARY:
Stress is known to trigger acute pain crisis of sickle cell disease (SCD). SCD is an inherited blood disorder that afflicts about 100,000 people in the United States, and is among the most common lethal genetic diseases in the United States. Though worldwide in distribution, in the US it is most commonly found in African Americans. Its best known complication is severe, recurrent relentless pain, often known as pain crisis. Non-drug treatment for SCD pain such as cognitive coping interventions have been shown to be effective for reducing SCD pain intensity, but they are complicated, multifaceted, and time-consuming. A simple and cost-effective alternative such as guided imagery (GI) could reduce the effect of stress on SCD pain. GI is an intervention where patients listen to and view audio-visual recordings while being directed to visualize themselves being immersed in that scene or scenario. There are no published studies on the use of GI as a simple stress coping intervention or tracking stress in a systematic manner as a trigger for SCD pain.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age or older,
* Diagnosis of SCD,
* Self-reported pain of at least 3 on a 0-10 scale related to SCD,
* Spoke and read English, and
* Self-identified as being of African or Hispanic descent.

Exclusion Criteria:

* Legally blind or physically unable to complete procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-11; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Current stress | Immediate (baseline)
  Stress intensity scale: A 3-item scale that asks patients to report their current, least, and worst stress intensity today, on a scale of 0 to 10, where 0 is "no stress" and 10 is "stress as bad as it could be." We estimated intervention effects using linear regression with bootstrapping.
Current pain | Immediate (baseline)
  PAINReportIt® Pain intensity scale: A 3-item scale that asks patients to report their current, least, and worst pain intensity today, on a scale of 0 to 10, where 0 is "no pain" and 10 is "pain as bad as it could be." We estimated intervention effects using linear regression with bootstrapping.
Average stress intensity | Short-term (2 weeks)
  Stress intensity scale: A 3-item scale that asks patients to report their current, least, and worst stress intensity today, on a scale of 0 to 10, where 0 is "no stress" and 10 is "stress as bad as it could be." We averaged the three scores to create an average stress intensity score. We estimated intervention effects using linear regression with bootstrapping.
Composite pain index | Short-term (2 weeks)
  PAINReportIt® Composite pain index (CPI): A a multidimensional representation of pain calculated by averaging the individual proportional scores for each of the four pain dimensions: (1) number of pain sites; (2) pain intensity; (3) total pain rating index (from the McGill Pain Questionnaire [MPQ], pain quality); and (4) pain pattern score. the scores for the CPI range from 0 to 100. We estimated intervention effects using linear regression with bootstrapping.

CONTACTS AND LOCATIONS:
Overall Officials: Miriam O Ezenwa, PhD, RN, Principal Investigator — University of Illinois at Chicago

REFERENCES:
- [Derived] Ezenwa MO, Yao Y, Engeland CG, Molokie RE, Wang ZJ, Suarez ML, Wilkie DJ. A randomized controlled pilot study feasibility of a tablet-based guided audio-visual relaxation intervention for reducing stress and pain in adults with sickle cell disease. J Adv Nurs. 2016 Jun;72(6):1452-63. doi: 10.1111/jan.12895. Epub 2016 Jan 15. PMID 26768753